CLINICAL TRIAL: NCT02051855
Title: NeoAdapt 2: An Observational Study Investigating Novel Biomarkers in the Evaluation and Treatment of Neonatal Circulatory Insufficiency in Infants Older Than 33 Weeks Gestational Age
Brief Title: NeoAdapt 2: An Observational Study Investigating Novel Biomarkers in the Evaluation and Treatment of Neonatal Circulatory Insufficiency
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Dr Liam Mahoney, Clinical Research Fellow in Paediatrics, Brighton and Sussex University Hospitals NHS Trust
Other Study IDs: IRAS: 145205
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Circulatory Failure
Keywords: Neonates; Superior Vena Cava Flow; Pleth Variability Index; Dobutamine; Intensive Care
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Two blood samples of 400µl each will be obtained for each infant receiving dobutamine.
  Samples for the pharmacokinetic studies will utilise micro assays to minimise the amount of blood taken and will coincide with the taking of clinically indicated sample to reduce the burden placed on neonates included in this study.
Oversight: Data Monitoring Committee: No

SUMMARY:
Circulatory failure can affect up to 50% of premature infants that are admitted to neonatal intensive care. This can be because their heart muscle is not developed enough to send blood to vital organs such as the brain. This can lead to severe short term problems such as kidney failure and contribute to poor long term development such as cerebral palsy. In addition babies born too early may need more time to adapt from a circulation that relies on the placenta in the womb to one that is self sufficient.

Doctors need to be able to accurately measure the blood supply in an infant. However there is no agreement on how best to do this. This makes decisions about when to treat an infant difficult. Doctors may use drugs such as dopamine or dobutamine to help a babies circulation. However these drugs have not been tested properly in babies older than 33 weeks gestation.

This study proposes to observe the way babies older than 33 weeks circulatory problems are treated in the first three days of life. In addition the study will look at two new measurements of a babies blood supply to see if they are a better measure of when an infant needs treatment. This will involve an ultrasound scan of the heart and measurement of the child's oxygen levels from a probe placed on their hand or leg. The study will also look at how the drug dobutamine is processed by babies. This will be done from two small extra blood tests. The aim of the study is to help clinicians refine the identification and treatment of circulatory failure in premature babies.

DETAILED DESCRIPTION:
Research has shown that there is large difference in how doctors treat this circulatory failure. This is because there is no agreed definition for this condition. By investigating new methods of assessing a babies circulatory status we intend to help create a new definition of circulatory failure which will in turn help doctors create further studies to identify infants with circulatory failure and find the best ways of treating this condition in babies. So far research in this area has been confined to babies born at less than 33 weeks gestation. We intend to extend the knowledge in the area to infants older that 33 weeks gestation.

Dobutamine is a drug that does not have a license for use in premature infants. In the future all new drugs will need to be studied in children before a license for them is given. In addition the European Community are encouraging that research is undertaken to look into the use of old drugs which are used in babies. As mentioned previously there is very little data to show how dobutamine is handled by babies and this study will contribute to new information on how this drug should be given to babies safely.

This is a pilot observational study in infants older than 33 weeks gestational age. The population will be observed for the diagnostic measures used to trigger treatment for circulatory failure. Treatment decisions will be made according to the preference of the responsible doctors. The treatment decision will be documented by the research team and the effect of that treatment on diagnostic measures will be recorded.

There will be an additional sub study involving those infants who receive dobutamine. This study will look at how the babies handle this drug.

WHAT WILL HAPPEN TO RESEARCH PARTICIPANTS

Infants will receive the same care as any other infant admitted to the neonatal intensive care unit. If the attending medical team decide that the infant is suffering from circulatory failure then they will receive treatment in the same way as other babies not involved in the study would. This may involve the giving of fluid through a vein, or the use of drugs such as dobutamine.

All infants who are admitted to neonatal intensive care unit will have all the standard tests and observations that infants would have. For babies included in the study for the first three days of their lives all included infants will have two specific measurements once a day. These are known as:-

1. Superior vena cava flow assessment- This involves measuring the blood flow through one of large veins that is connected to the babies' heart using an ultrasound machine. It is a painless procedure that is well tolerated by infants.
2. Pleth variability index- This involves placing a small probe on the baby's hand or foot that will measure their oxygen levels. This will be done at the same time as the superior vena cava flow assessment is performed. Again this is a painless procedure that is well tolerated by infants.

The study will also record important relevant outcomes of routine tests performed on infants admitted other neonatal unit:

1. Brain ultrasound appearances during their stay on the unit.
2. Monitoring of clinical parameters, observations and laboratory tests.
3. Major clinical diagnoses.

If an infant receives dobutamine then they will have two small blood samples taken to investigate how drug is processed in babies. This will be done via methods that minimise pain and distress for the infants involved in the study.

This will be an observational pilot cohort study with the aim of improving the definition of circulatory failure in neonates and document current treatment strategies for haemodynamic insufficiency during the transitional circulation in infants greater than 33 weeks gestational age who are admitted to the neonatal unit (NICU) for intensive care.

Inclusion criteria will be

1. Neonates >33 weeks gestational age admitted to the neonatal intensive care unit
2. Postnatal age <72 hours;
3. Parental informed consent; This population will be observed with regard to which diagnostic measures lead to treatment decisions and what the effect of those decisions are on the various diagnostic measures. Decision-making for their treatment will be based on clinical guidelines in operation at Trevor Mann Bay Unit and clinician preference.

The assessment of SVC flow and PVI will only be done in every 24 hours for the first 72 hours of life in babies.

Primary Outcome Measure Values for SVCF and PVI in neonates aged older than 33 weeks gestational age receiving intensive care derived from Echo-D and plethysmographic studies .

Observed Clinical Outcome Measures

Cranial US appearances

The analysis of the findings on cranial ultrasound scan will be interpreted in the light of a baseline scan, to be performed as soon as possible after birth on enrolment, to avoid ascribing the effect of antenatal insults to postnatal events.

Treatments for Circulatory Failure Infants will receive treatment according to the preference of the responsible physician. As is common practice, dobutamine, dopamine and/or other treatments (including other cardiovascular drugs and/or volume replacement therapy with normal saline) will be administered.

Dose of administration The dose of administration of dobutamine will be at the discretion of the responsible physician. We envisage that dobutamine will typically be started between 2.5 and 5 mcg/kg/min and increased in steps of 5 mcg/kg/min to a maximum of 20 mcg/kg/min with a given time frequency if no response is seen.

Any changes to the treatment strategy will be documented by the responsible physician.

Criteria for Up-Titration of Medication Dose escalation will be guided by clinical judgment. Clinicians will be asked to record the criteria they used in order to make this decision.

Criteria for Down-Titration Dose reduction will be guided by clinical judgment. Clinicians will be asked to record the criteria they used in order to make this decision.

Further treatment If there is no response to dobutamine at 20 mcgg/k/min or the clinical response is considered by the attending physician to be inadequate, further treatment will be at the discretion of the attending physician who will be asked to record the reasons for the change in treatment strategy as well as the additional treatment that is given to the patient.

Concomitant therapy There will be no per-protocol concomitant medication or treatment. Accordingly, other important co-interventions will follow specific centre protocols and will be recorded in the case record form.

PHARMACOKINETICS (PK) SUB-STUDY

Aim of the PK sub-studies The aim of the sub-study is to give preliminary information in order to try and construct a population PK model. Given the uncertainties regarding the PK of dobutamine in infants receiving intensive care we shall assess its elimination half life. This is defined as the amount of time for the quantity of a concentration to fall by half.

Half-life sub-study We will perform a preliminary study on all the infants included in NeoAdapt 2 that receive dobutamine as treatment for haemodynamic insufficiency. Two blood samples, of 400 μl each, will be obtained from each of these patients. The first sample will be drawn after the end of the infusion, at the time when dobutamine ceases reaching the systemic circulation of the neonate, defined as time end (te).

The second sample will be taken at different study time points after the end of infusion:

5 min after te 15 min after te 45 min after te 2 hours after te 6 hours after te Two infants will be allocated to each time point. Sampling times will be assigned randomly to the patients.

Plasma samples will be sent to the laboratory for the quantification of dobutamine.

ELIGIBILITY:
Inclusion Criteria:

* Neonates >33 weeks gestational age
* Postnatal age <72 hours
* Parental informed consent
* Admitted to the neonatal intensive care unit

Exclusion Criteria:

* Non-viability
* Congenital hydrops or malformations likely to affect cardiovascular adaptation
* Surgery planned within 72 hours of birth
* Chromosomal anomalies
* Informed consent form (ICF) not signed

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged older than 33 weeks gestational admitted to the neonatal intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Superior Vena Cava Flow (SVCF) in infants older than 33 weeks gestational age receiving intensive care | Once a day for a maximum of three days after birth
  After consent and enrolment, Echo-D will be performed as soon possible in the first 24 hours a babies life. Echo-D assessments will be repeated every 24 hours during the first 72 hours of postnatal life, whenever possible. This in this measurement over the first three days of life will be recorded.
Pleth Variability Index (PVI) in infants older than 33 weeks gestational age receiving intensive care | Once a day for a maximum of three days after birth
  After consent and enrolment, PVI will be performed as soon possible in the first 24 hours a babies life. PVI assessments will be repeated every 24 hours during the first 72 hours of postnatal life, whenever possible. The change in this measurement in the first three days of life will be recorded
Pharmacokinetic data for the elimination half life of dobutamine when it is used for circulatory failure in infants older than 33 weeks gestational age. | If dobutamine is given to an infant in the first three days of life
  If dobutamine is given to an infant in the first three days of life 2 blood samples will be taken for pharmacokinetic analysis of dobutamine to determine its elimination half life.

SECONDARY OUTCOMES:
SVCF and PVI values correlation to each other and to parameters that assess circulatory status such as mean blood pressure and capillary refill time | Over the first 3 days of life
  Correlation analysis will be used to determine if there is an association between SVCF and PVI values to common parameters that are used in the neonatal intensive care setting to assess the haemodynamic status of an infant.
SVCF and PVI values relationship to clinical outcomes | Over the first three days of life
  Clinical outcomes for infants who are suffering from hypoxic ischemic encephalopathy, such as cranial ultrasound appearances, will be recorded. These outcomes will be compared to the SVCF and PVI values gained to see if either measurement is predictive of such clinical outcomes.
SVCF and PVI values and dobutamine treatment for circulatory failure | Over the first three days of life
  Comparisons between the will be made between SVCF and PVI values gained from infants who were and those who were not receiving dobutamine at the time of these measurements to see if there is a significant difference between the values gained.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Mahoney, BMBS, MRCPCH, Principal Investigator — Brighton & Sussex Medical School/Brighton & Sussex Universitys NHS Trust
Locations (1):
- Trevor Mann Baby Unit, Brighton, Sussex, United Kingdom

REFERENCES:
- See also: This is the main clinical trial the study is associated with — http://neocirculation.eu/